CLINICAL TRIAL: NCT04712981
Title: Adapting the HOPE Online Support Intervention to Increase MAT Uptake Among OUD Patients
Brief Title: Adapting the HOPE Online Support Intervention to Increase Uptake of Medications for Opioid Use Disorder
Acronym: HOPE MOUD
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Irvine (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Sean D Young, Professor, University of California, Irvine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20205625; 4R33AT010606 (NIH)
Record Dates: First submitted 2021-01-11; First posted 2021-01-19 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-08

CONDITIONS: Opioid-use Disorder
Keywords: online community
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): HOPE intervention peer-led online community
  Interventions: Behavioral: HOPE
- Control (No Intervention): Online community without HOPE intervention psychological components

INTERVENTIONS:
Behavioral: HOPE — Peer leaders/role models will be trained in HOPE intervention fundamentals and assigned to online community groups with participants.
  Arms: Intervention

SUMMARY:
In a randomized controlled trial, with 3, 6-month and 1-year follow-up, this application aims to explore whether and how the HOPE intervention can be adapted to increase MOUD uptake among OUD patients, assess the effectiveness of using HOPE to increase MOUD requests, and analyze online community data to improve future intervention implementation and sustainability.

DETAILED DESCRIPTION:
The proposed study is a low-risk, randomized control trial to assess the efficacy of the HOPE (Harnessing Online Peer Education) intervention, an evidenced-based peer-led social media/online community intervention (e.g., Facebook Groups), to increase self-reported requests for medications for opioid use disorder (MOUD) among patients with moderate to severe opioid use disorder (OUD). Participants will be recruited using a variety of recruitment methods including social media sites (e.g., Facebook), referral by physicians, medical records, research study websites (e.g., UCIMC Clinical Trials website), and study flyers disseminated at various venues, including clinics, group meetings, and shelters. Once enrolled, participants will be randomly assigned to an intervention or control group. Intervention group participants will be invited to join a private and hidden (unable to be viewed or searched for by others) group on Facebook, with approximately 6 peer leaders included in the group. Those in the control group will be invited into a Facebook group, but without peer leaders. The intervention will last 12 weeks. Study measures will be collected at the beginning of the study (baseline), after the completion of the intervention (3 months), with follow up surveys at 6 and 12 months after the study.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years of age;
2. Resident of CA, NV, AZ, OR, WA;
3. English speakers only;
4. Has moderate to severe OUD;
5. Is not currently prescribed MOUD;
6. Reports using social media at least 2x per week;
7. Has, or is willing to create a Facebook/social media account and accept a friend request and group invite from our study social media page

Exclusion Criteria

1. Anyone who does not fit inclusion criteria above
2. Was a participant in phase I of the study
3. Participants with active, unstable opioid, alcohol, sedative, or other substance use and/or unstable medical or psychiatric conditions as assessed by the study questionnaires will be reviewed by the study physician consultants and will be excluded and referred for acute care including detoxification, if needed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 640 (Actual)
Dates: Start 2021-04-29 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Number of requests to receive a resource on medications that can be used to treat opioid use disorder | request during the course of the 12-week community
  Participants will be invited to request an informational resource on medications for opioid use disorder as well as to ask for assistance scheduling an appointment with a provider on this topic. We will count the number of participants making this request

CONTACTS AND LOCATIONS:
Overall Officials: Sean D Young, PhD, Principal Investigator — University of California, Irvine
Locations (1):
- University of California, Irvine, Irvine, California, United States

IPD SHARING:
Plan to Share IPD: No